CLINICAL TRIAL: NCT01642043
Title: Point-of-Care Ultrasound in Greater Trochanteric Pain Syndrome (GTPS)
Brief Title: Point-of-Care Ultrasound in Greater Trochanteric Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Minna Jean Kohler, Director, Musculoskeletal Ultrasound- Division of Rheumatology, Allergy, and Immunology, Massachusetts General Hospital
Other Study IDs: 2012p001126
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Greater Trochanteric Pain Syndrome
Keywords: greater trochanteric pain syndrome; trochanteric bursitis; lateral hip pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Greater trochanteric pain syndrome (GTPS) is a common cause of musculoskeletal pain.

The primary aim of this study is to describe the soft tissue and bony structural ultrasound (US) findings identified in the lateral hip and iliotibial band (ITB) in patients presenting with greater trochanteric pain syndrome (GTPS) in an outpatient rheumatology clinic.

DETAILED DESCRIPTION:
GTPS, widely known as trochanteric bursitis, encompasses a spectrum of disorders (gluteal tendinopathy, tears, bursitis, and ITB syndrome) that are difficult to distinguish by clinical exam alone. Better understanding of US imaging characteristics in relation to clinical symptoms may be helpful in identifying those patients who would most benefit from corticosteroid injections and other non-operative treatment options.

Point-of-care musculoskeletal US use has been shown to reduce repeated hospital appointments, improve accuracy of diagnosis, and provide expedited treatment, thus improving quality of care in an outpatient musculoskeletal clinic. US assessment is not routinely included in the management of GTPS patients and ideal imaging modalities are not established.

ELIGIBILITY:
Inclusion Criteria:

* Lateral hip pain thought to be due to GTPS as evidenced by tenderness to palpation of the lateral hip over the greater trochanter
* Have a pain score of at least 2 out of 10 on an 11-point numeric rating scale
* Lateral hip pain for at least 1 week
* For participants with bilateral GTPS, the most symptomatic hip will be considered the study hip
* Have a telephone

Exclusion Criteria:

* Inability to give informed consent
* BMI > 40
* Evidence of severe OA of the study hip by X-ray
* Avascular necrosis of the study hip
* Groin pain at rest or with log-rolling
* Hip internal rotation range of motion < 15 degrees
* Prior fracture involving the study hip or femur
* Prior hip surgery or prosthesis in the painful hip
* Paralysis or paresis of the lower extremity
* Wheelchair bound
* Open wound or skin lesions in the lateral hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient rheumatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Descriptive diagnostic ultrasound findings of the bony and soft tissue structures of the lateral hip and iliotibial band | Baseline
  Presence of tendinopathy, tendon tears, bursitis, enthesophytes, calcifications

SECONDARY OUTCOMES:
Pain with rest measured by a numeric rating scale | Baseline and 2 weeks
Pain with activity as measured by a numeric rating scale | Baseline and 2 weeks
Demographics- composite | Baseline
  age, gender, race/ethnicity, education, occupation, comorbidities, overall health status.
Pressure point threshold as measured by an algometer | Baseline
Clinical data: Predictors of treatment response- composite | Baseline
  * Duration of pain
  * Body Mass Index
  * Physical exam findings
  * Treatments tried in the past
  * Presence of back pain

CONTACTS AND LOCATIONS:
Overall Officials: Minna J. Kohler, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States